CLINICAL TRIAL: NCT06296004
Title: Relation Between Nail Fold Capillaroscopy, Optical Coherence Tomography Angiography, and Femoral Vein Wall Thickness in Behçet's Disease
Brief Title: Relation Between Nail Fold Capillaroscopy, Optical Coherence Tomography Angiography, and Femoral Vein Wall Thickness in Behçet's Disease Relation Between Nail Fold Capillaroscopy, Optical Coherence Tomography Angiography, and Femoral Vein Wall Thickness in Behçet's Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Elzahraa Awny Fathy, Assistant lecturer, Assiut University
Other Study IDs: CAPILLAROSCOPY behcet disease
Record Dates: First submitted 2024-02-21; First posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-02

CONDITIONS: Behçet's Disease
MeSH Terms: conditions — Behcet Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- adult patient with Behçet's Disease: . Adult BD patients who fulfilling the criteria for the diagnosis by International Team for the Revision of the International Criteria for Bechet's Disease .
  Interventions: Device: Nail Fold Capillaroscopy, Optical Coherence Tomography Angiography, and Femoral Vein Wall Thickness by U.S
- healthy subjects: apparently healthy subjects
  Interventions: Device: Nail Fold Capillaroscopy, Optical Coherence Tomography Angiography, and Femoral Vein Wall Thickness by U.S

INTERVENTIONS:
Device: Nail Fold Capillaroscopy, Optical Coherence Tomography Angiography, and Femoral Vein Wall Thickness by U.S — Complete blood count (CBC) Erythrocyte sedimentation rate (ESR) measured by standard westergren method (mm/h).
  Serum C-reactive protein (CRP) Liver function tests: aspartate transaminase (AST), alanine transaminase (ALT), serum albumin, serum bilirubin.
  Renal function tests: serum creatinine and blood urea. Complete urine analysis.
  Optical coherence tomography angiography (OCTA): . Bilateral common femoral vein (CFV) Doppler US

SUMMARY:
Relation between Nail Fold Capillaroscopy, Optical Coherence Tomography Angiography, and Femoral Vein Wall Thickness in Behçet's Disease

DETAILED DESCRIPTION:
Behçet disease (BD) is a multisystemic, autoinflammatory, chronic illness that is quite common in the nations along the ancient Silk Road. It is characterized by immune-mediated vasculitis, which can affect blood vessels of any size throughout all organ systems Vascular involvement, is one of the more serious symptoms of BD, which is considered to have a poor prognostic value. The majority of research on vascular involvement in BD focuses on large vessel involvement; however, less research discusses microvascular damage. Capillaroscopy is a non-invasive diagnostic method used to assess small vessels in the microcirculation Furthermore, ocular inflammation is the most prevalent form affecting more than 70% of Behçet diseased patients in the form of relapsing, remitting uveitis Fluorescein angiography is currently the gold standard for documenting and tracking posterior segment involvement in BD because it can easily detects retinal ischemia, macular edema, and retinal vascular leakage . Nevertheless, this process is invasive, necessitating the injection of an external dye, and its depth resolution is restricted Recently, optical coherence tomography angiography (OCT-A) has emerged as a highly effective method for obtaining high resolution en face images of the choroidal and retinal microvasculature, as well as for analyzing changes in the choriocapillaris, deep capillary plexus, and superficial capillary plexus independently . OCT-A allows for the assessment of both qualitative and quantitative alterations within the retinal microvasculature. Few research have looked into the use of OCT-A in Behçet uveitis, despite the fact that its role in the evaluation of retinal vascular diseases, such as diabetic retinopathy, retinal venous occlusions, retinal arterial occlusions, and age-related macular degeneration, has been thoroughly examined in the recent literature It has recently been proposed that venous wall thickness (VWT), measured by Doppler ultrasonography (US), can serve as an indirect sonographic marker for the extent of vascular end organ damage, including venous illness. Increased VWT, particularly in the femoral and popliteal veins, has been shown in numerous investigations to be a highly significant clinical characteristic in BD However, whether US findings are correlated with vascular involvement in BD is still unknown. It has been determined that the most suitable site to evaluate VWT using US is the common femoral vein (CFV). A sensitivity of 81-22% and a specificity of 78.4-81.1.1% have been reported for the VWT cut-off point of ≥0.5 mm in the diagnosis of BD. It has therefore been suggested as an efficient and non-invasive method for diagnosing BD

ELIGIBILITY:
Inclusion Criteria:

1. Adult BD patients who fulfilling the criteria for the diagnosis by International Team for the Revision of the International Criteria for Bechet's Disease .
2. Accept to participate in the current study -

Exclusion Criteria:

1. Individuals with other autoimmune diseases (rheumatoid arthritis dermatomyositis, scleroderma, mixed connective tissue disease).
2. Patients with high myopia or media opacities preventing high-quality imaging like cataract and cornea guttata, vitreoretinal disease, previous retinal surgery, macular edema, glaucoma or neurological disease.
3. Patients with other comorbidities as diabetes, hypertension were excluded from the study.
4. Refused to participate in the current study.

   -

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study will include 80 participants:
  Group 1: 40 patients with who fulfilling the criteria for the diagnosis by International Team for the Revision of the International Criteria for Bechet's Disease (Disease et al., 2014).
  . Group 2: 40 healthy matched controls.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
measuring parameter of Nail Fold Capillaroscopy in behcet disease | 1 year
  using previous parameters in diagnosis of vascular affection in behcet disease
measuring parameter of Optical Coherence Tomography Angiography in behcet disease | 1 year
  using previous parameters in diagnosis of vascular affection in behcet disease
measuring parameter of Femoral Vein Wall Thickness in behcet disease | 1year
  using previous parameters in diagnosis of vascular affection in behcet disease

SECONDARY OUTCOMES:
relation between Nail Fold Capillaroscopy and activity of behcet disease | 1 years
  using previous parameters in measuring disease activity
relation between Optical Coherence Tomography Angiography and activity of behcet disease | 1 year
  using previous parameters in measuring disease activity
relation between Femoral Vein Wall Thickness and activity of behcet disease | 1 year
  using previous parameters in measuring disease activity

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alibaz-Oner F, Ergelen R, Yildiz Y, Aldag M, Yazici A, Cefle A, Koc E, Artim Esen B, Mumcu G, Ergun T, Direskeneli H. Femoral vein wall thickness measurement: A new diagnostic tool for Behcet's disease. Rheumatology (Oxford). 2021 Jan 5;60(1):288-296. doi: 10.1093/rheumatology/keaa264. PMID 32756998
- [Background] Alibaz-Oner F, Direskeneli H. Assessment of venous wall thickness with Doppler ultrasonography may be a diagnostic tool for Behcet's disease. Int J Rheum Dis. 2019 May;22(5):767-768. doi: 10.1111/1756-185X.13574. No abstract available. PMID 31062939
- [Background] Alten F, Heiduschka P, Clemens CR, Eter N. Exploring choriocapillaris under reticular pseudodrusen using OCT-Angiography. Graefes Arch Clin Exp Ophthalmol. 2016 Nov;254(11):2165-2173. doi: 10.1007/s00417-016-3375-1. Epub 2016 May 18. PMID 27193430
- [Background] Bhakta BB, Brennan P, James TE, Chamberlain MA, Noble BA, Silman AJ. Behcet's disease: evaluation of a new instrument to measure clinical activity. Rheumatology (Oxford). 1999 Aug;38(8):728-33. doi: 10.1093/rheumatology/38.8.728. PMID 10501420
- [Background] Bonini Filho MA, Adhi M, de Carlo TE, Ferrara D, Baumal CR, Witkin AJ, Reichel E, Kuehlewein L, Sadda SR, Sarraf D, Duker JS, Waheed NK. OPTICAL COHERENCE TOMOGRAPHY ANGIOGRAPHY IN RETINAL ARTERY OCCLUSION. Retina. 2015 Nov;35(11):2339-46. doi: 10.1097/IAE.0000000000000850. PMID 26457398
- [Background] Cheng D, Shen M, Zhuang X, Lin D, Dai M, Chen S, Lu F, Wang Y. Inner Retinal Microvasculature Damage Correlates With Outer Retinal Disruption During Remission in Behcet's Posterior Uveitis by Optical Coherence Tomography Angiography. Invest Ophthalmol Vis Sci. 2018 Mar 1;59(3):1295-1304. doi: 10.1167/iovs.17-23113. PMID 29625452
- [Background] Chojnowski MM, Felis-Giemza A, Olesinska M. Capillaroscopy - a role in modern rheumatology. Reumatologia. 2016;54(2):67-72. doi: 10.5114/reum.2016.60215. Epub 2016 Jun 3. PMID 27407282
- [Background] de Carlo TE, Romano A, Waheed NK, Duker JS. A review of optical coherence tomography angiography (OCTA). Int J Retina Vitreous. 2015 Apr 15;1:5. doi: 10.1186/s40942-015-0005-8. eCollection 2015. PMID 27847598
- [Background] International Team for the Revision of the International Criteria for Behcet's Disease (ITR-ICBD). The International Criteria for Behcet's Disease (ICBD): a collaborative study of 27 countries on the sensitivity and specificity of the new criteria. J Eur Acad Dermatol Venereol. 2014 Mar;28(3):338-47. doi: 10.1111/jdv.12107. Epub 2013 Feb 26. PMID 23441863
- [Background] Khairallah M, Abroug N, Khochtali S, Mahmoud A, Jelliti B, Coscas G, Lupidi M, Kahloun R, Ben Yahia S. OPTICAL COHERENCE TOMOGRAPHY ANGIOGRAPHY IN PATIENTS WITH BEHCET UVEITIS. Retina. 2017 Sep;37(9):1678-1691. doi: 10.1097/IAE.0000000000001418. PMID 28002270
- [Background] Lupidi M, Cerquaglia A, Chhablani J, Fiore T, Singh SR, Cardillo Piccolino F, Corbucci R, Coscas F, Coscas G, Cagini C. Optical coherence tomography angiography in age-related macular degeneration: The game changer. Eur J Ophthalmol. 2018 Jul;28(4):349-357. doi: 10.1177/1120672118766807. Epub 2018 Apr 6. PMID 29623720
- [Background] • Onan, D., Uysal, P., Hayran, Y., Şahin Dalgıç, G., Hayran, M., Artüz, F. & Yalçin, B. (2019) Dermatoscopic Assessment of Nailfold Capillary Abnormalities in Behçet's Disease and Correlation of the Findings with Disease Activity and Severity. Dermatologica Sinica, 37, 40-45.
- [Background] Samara WA, Shahlaee A, Adam MK, Khan MA, Chiang A, Maguire JI, Hsu J, Ho AC. Quantification of Diabetic Macular Ischemia Using Optical Coherence Tomography Angiography and Its Relationship with Visual Acuity. Ophthalmology. 2017 Feb;124(2):235-244. doi: 10.1016/j.ophtha.2016.10.008. Epub 2016 Nov 23. PMID 27887743
- [Background] Samara WA, Shahlaee A, Sridhar J, Khan MA, Ho AC, Hsu J. Quantitative Optical Coherence Tomography Angiography Features and Visual Function in Eyes With Branch Retinal Vein Occlusion. Am J Ophthalmol. 2016 Jun;166:76-83. doi: 10.1016/j.ajo.2016.03.033. Epub 2016 Mar 31. PMID 27038893
- [Background] Sambhav K, Grover S, Chalam KV. The application of optical coherence tomography angiography in retinal diseases. Surv Ophthalmol. 2017 Nov-Dec;62(6):838-866. doi: 10.1016/j.survophthal.2017.05.006. Epub 2017 Jun 1. PMID 28579550
- [Background] Somkijrungroj T, Vongkulsiri S, Kongwattananon W, Chotcomwongse P, Luangpitakchumpol S, Jaisuekul K. Assessment of Vascular Change Using Swept-Source Optical Coherence Tomography Angiography: A New Theory Explains Central Visual Loss in Behcet's Disease. J Ophthalmol. 2017;2017:2180723. doi: 10.1155/2017/2180723. Epub 2017 May 9. PMID 28596917
- [Background] Spaide RF, Fujimoto JG, Waheed NK, Sadda SR, Staurenghi G. Optical coherence tomography angiography. Prog Retin Eye Res. 2018 May;64:1-55. doi: 10.1016/j.preteyeres.2017.11.003. Epub 2017 Dec 8. PMID 29229445
- [Background] Tugal-Tutkun I, Ozdal PC, Oray M, Onal S. Review for Diagnostics of the Year: Multimodal Imaging in Behcet Uveitis. Ocul Immunol Inflamm. 2017 Feb;25(1):7-19. doi: 10.1080/09273948.2016.1205100. Epub 2016 Aug 19. PMID 27541278
- [Background] Yilmaz PT, Ozdemir EY, Alp MN. Optical coherence tomography angiography findings in patients with ocular and non-ocular Behcet disease. Arq Bras Oftalmol. 2021 May-Jun;84(3):235-240. doi: 10.5935/0004-2749.20210031. PMID 33567020